CLINICAL TRIAL: NCT04213170
Title: Prospective Phase II Clinical Study of Sintilimab Combined With Bevacizumab for Driving Gene-negative, Asymptomatic Brain Metastases From Non-small Cell Lung Cancer
Brief Title: Sintilimab Combined With Bevacizumab for Brain Metastases From Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li-kun Chen, medical doctor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2019-050-01
Record Dates: First submitted 2019-12-25; First posted 2019-12-30 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-05

CONDITIONS: Brain Metastases; Non Small Cell Lung Cancer; Sintilimab; Bevacizumab
MeSH Terms: conditions — Brain Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — sintilimab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sintilimab and Bevacizumab (Experimental): Sintilimab 200mg d1 and Bevacizumab 15mg/kg d1 every 21 days
  Interventions: Drug: sintilimab

INTERVENTIONS:
Drug: sintilimab — Sintilimab 200mg d1 and Bevacizumab 15mg/kg d1 q21d
  Other Names: bevacizumab

SUMMARY:
This is a prospective phase II clinical study to assess the efficacy of Sintilimab combined with Bevacizumab for driving gene-negative, asymptomatic brain metastases from non-small cell lung cancer by intracranial ORR(iORR),also iPFS,ORR and PFS.The safety and tolerability is evaluated as well.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with NSCLC confirmed by histology or cytology;
2. Patients with asymptomatic brain metastasis or brain metastasis whose symptoms of intracranial hypertension have been alleviated after dehydration treatment should keep the clinical stable state for at least 2 weeks.For patients requiring hormone dehydration therapy, hormone therapy should be discontinued 3 days before the first dose of the study drug.
3. Appraisable disease, the diameter of at least one measurable lesion in the brain must be 5mm;
4. The detection results of tumor tissue biomarkers should meet the following conditions simultaneously: EGFR has no sensitive mutation;ALK rearrangement negative;for never treated patients, they also needed to meet PD-L1 >50% or TMB>12Mut/Mb (second-generation sequencing).
5. Adult patients (≥ 18 years and ≤75 years). ECOG Performance Status 0 or 1 Life expectancy of at least 12 weeks.,Haemoglobin ³ 10.0 g/dl, Absolute neutrophil count (ANC) ³1.5 x 109/L, platelets ³ 100 x 109/L. Total bilirubin £ 1.5 x upper limit of normal (ULN). ALT and AST < 2.5 x ULN in the absence of liver metastases, or < 5 x ULN in case of liver metastases. Creatinine clearance ³ 60ml/min (calculated according to Cockcroft-gault formula).
6. Ability to follow study and follow-up procedures;
7. Prior to the implementation of any trial-related procedures, a written informed consent shall be signed.

Exclusion Criteria:

1. Mixed non-small cell and small cell carcinoma;
2. Brain metastasis with hemorrhage;
3. Currently participating in interventional clinical research and treatment, or receiving other research drugs or using research instruments within 4 weeks before the first dose;
4. Previously received the following therapies: anti-PD-1, anti-PD-L1 or anti-PD-L2 drugs or drugs targeting another stimulation or synergistic inhibition of T cell receptors (e.g., CTLA-4, CD137);
5. Received solid organ or blood system transplantation;
6. Received >30GY pulmonary radiotherapy 6 months before the first dose;
7. Active autoimmune diseases requiring systemic treatment (such as the use of disease-relieving drugs, corticosteroids or immunosuppressants) occurred within 2 years before the first dose.Alternative therapies (such as thyroxine, insulin, or physiological corticosteroids for adrenal or pituitary insufficiency) are not considered systemic;
8. Received systemic glucocorticoid therapy or any other form of immunosuppressive therapy within 7 days before the first dose of the study or diagnosed as immunodeficiency;a physiological dose of glucocorticoid (10 mg/ day of prednisone or equivalent) is permitted;
9. History of non-infectious pneumonia requiring glucocorticoid therapy or current interstitial pulmonary disease was found within 1 year before the first dose;
10. History of human immunodeficiency virus (HIV) infection (i.e. HIV 1/2 antibody positive)
11. Untreated active hepatitis;
12. History of hemoptysis within 3 months prior to selection, that is, at least 1/2 teaspoon of blood was coughed up;
13. Imaging showed signs of tumor invasion into the great vessels.The investigator or radiologist must rule out patients whose tumors have completely approached, wrapped, or invaded the intravascular space of the great vessels
14. Serious uncontrolled coagulation disorder or thrombi-embolic complications within 6 months prior to study start or history of serious bleeding complications.
15. Major surgical procedures within 4 weeks prior to study entry.
16. Minor surgery, including insertion of an indwelling catheter, within 24 hours prior to the first bevacizumab infusion.
17. Non-healing wound, active peptic ulcer or bone fracture.
18. History of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 6 months of enrollment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-04-29 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
iORR | 3.5 years
  intracranial objective response rate

SECONDARY OUTCOMES:
iPFS | 3.5 yesrs
  intracranial progression free survival
ORR | 3.5 years
  objective response rate
PFS | 3.5 years
  progression free survival

CONTACTS AND LOCATIONS:
Overall Officials: Likun Chen, doctor, Study Director — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University of Cancer Center, Guangzhou, Guangdong, China